CLINICAL TRIAL: NCT06854484
Title: AVEIR™ Leadless Pacemaker United Kingdom Registry
Brief Title: AVEIR™ Leadless Pacemaker (LP) United Kingdom (UK) Registry
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: AVEIR™ Registry; Medical Affairs CR24562 (Other Grant/Funding Number: Abbott Medical UK Ltd.)
Record Dates: First submitted 2025-01-28; First posted 2025-03-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Bradycardia; Atrio-Ventricular Block; Syncope
Keywords: AVEIR leadless pacemaker
MeSH Terms: conditions — Bradycardia; Syncope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients requiring leadless pacemaker insertion: Patients who require leadless pacemaker to manage their heart condition
  Interventions: Device: AVEIR™leadless pacemaker

INTERVENTIONS:
Device: AVEIR™leadless pacemaker — AVEIR™ leadless pacemaker implantation

SUMMARY:
This observational study will follow patients requiring implantation of leadless pacemaker for 5 years after implantation. The main goal is to evaluate the long term safety and efficacy of AVEIR™ leadless pacemaker device in the usual clinical settings within the UK National Health Service. In addition, the study will collect data to understand patient characteristics receiving this type of pacemaker.

DETAILED DESCRIPTION:
AVEIR™ stimulator (Abbott) obtained the approvals in July 2023 and started to be implanted in patients in Europe. As a leadless pacemaker, the AVEIR™ Leadless Pacemaker (LP) does not need a connector, pacing lead, or pulse generator pocket. The LP is delivered percutaneously via the femoral vein through an AVEIR™ Introducer and Delivery Catheter. AVEIR™ LP is intended to provide bradycardia pacing as a pulse generator with built-in battery and electrodes for implantation. The LP is intended to provide sensing of intrinsic cardiac signals and delivery of cardiac pacing therapy to the target treatment group.

The purpose of this study is to understand long term safety and performance characteristic of this device. In addition, the study will collect anonymous clinical data and characteristics of the patients chosen to be implanted with AVEIR™ leadless pacemaker in routine clinical practice in approved centres across the UK.

Six hundred patients will be recruited in up to 15 centres during 2 years recruitment period. They will be followed up for 5 years after implantation of the leadless pacemaker. Investigators will record their age, sex, medical history, indications for receiving AVEIR™ and any complications related to the implantation procedure or the device itself. All the data will be collected in an anonymous format. Patients will be followed up according to the standard of care in the national health care system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is intended to receive or was treated with a (AVEIR™) Leadless Transcatheter Pacing
2. Subject is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams; and
3. Subject has been informed of the nature of the study, agrees to its provisions, and has provided a signed written informed consent, approved by the Regional Ethics Committee (REC).

Exclusion Criteria:

1. Subject is not suitable for implantation of the leadless device according to the expert opinion of their cardiologist.
2. Subject is not willing to comply with clinical investigation procedures and does not agree to return for all required follow-up visits, tests, and exams
3. Subject has been informed of the nature of the study, but does not agree to its provisions, and has not provided a signed written informed consent, approved by the REC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive cardiology patients listed for leadless pacemaker implantation and fitted with AVEIR™ LP device in the usual clinical practice in the UK National Health Service centres.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients without complications related to the device or implantation procedure. | 5 years
  Complications arising from the procedure or the device will be recorded to evaluate the success rate of the implantation.
Percentage of patients requiring re-intervention. | 5 years
  Replacement, explant, upgrade, or modification of the position of the device are considered re-interventions which will be used to evaluate safety of the device.
Stimulation threshold (V) in the therapeutic zone | 5 years
  Minimum current needed to stimulate the paced chamber.
Percentage of stimulation in the therapeutic zone | 5 years
  Percentage of paced vs non paced heart beats.
Impedance (Ohm) of R waves in the therapeutic zone | 5 years
  Physiological measure recorded by the device.
Amplitudes of R waves (mV) in the therapeutic zone | 5 years
  Physiological measure recorded by the device.

SECONDARY OUTCOMES:
Age of patient (years) at AVEIR ™ leadless pacemaker implantation | 5 years
  Collected as part of the demographics data for the patient group under investigation.
Sex of patient at AVEIR ™ leadless pacemaker implantation | 5 years
  Collected as part of the demographics data for the patient group under investigation.
Medical history at AVEIR ™ leadless pacemaker implantation | 5 years
  List of significant cardiac or other comorbidities at the time of pacemaker implantation to describe patient population receiving AVEIR ™ leadless pacemaker.
Indications for AVEIR ™ leadless pacemaker implantation | 5 years
  Collected as part of the demographics data for the patient group under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wong, MD, Principal Investigator — Royal Brompton and Harefield Hospital
Locations (2):
- United Kingdom (2):
  - Royal Brompton Hospital, London, UK
  - The Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No